CLINICAL TRIAL: NCT00375401
Title: A 2-Year, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study To Evaluate The Long-Term Efficacy And Safety Of CP-945,598 In The Treatment Of Obese Subjects
Brief Title: A Long-Term Study To Examine The Effects Of CP-945,598 On Weight Loss And Safety
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5351025
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CP-945,598 Treatment A (Experimental)
  Interventions: Drug: CP-945,598 Treatment A
- CP-945,598 Treatment B (Experimental)
  Interventions: Drug: CP-945,598 Treatment B
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-945,598 Treatment A — Arm includes CP-945,598 Treatment A plus Dietary, Physical Activity, and Weight Loss Counseling
  Arms: CP-945,598 Treatment A
Drug: CP-945,598 Treatment B — Arm includes CP-945,598 Treatment B plus Dietary, Physical Activity, and Weight Loss Counseling
  Arms: CP-945,598 Treatment B
Drug: Placebo — Arm includes Placebo plus Dietary, Physical Activity, and Weight Loss Counseling
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the long-term weight loss and safety of CP-945,598 in obese adults

DETAILED DESCRIPTION:
The CP-945,598 program was terminated on November 3, 2008 due to changing regulatory perspectives on the risk/benefit profile of the CB1 class and likely new regulatory requirements for approval. No safety issues were involved in the termination decision.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults with a body mass index > or = 30 kg/m2; > or = to 27 kg/m2 for those with obesity-related comorbidities including hypertension and dyslipidemia

Exclusion Criteria:

* Pregnancy
* Diabetes
* Adults with serious or unstable current or past medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2536 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with 5% weight loss | 1 year
Change in body weight | 1 year

SECONDARY OUTCOMES:
Blood pressure, blood lipids and glucose, waist circumference, quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (75):
- United States (67):
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Waconia, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Olympia, Washington
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Oregon, Wisconsin
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351025&StudyName=A%20Long-Term%20Study%20To%20Examine%20The%20Effects%20Of%20CP-945%2C598%20On%20Weight%20Loss%20And%20Safety